CLINICAL TRIAL: NCT07155902
Title: Leveraging Community-to-facility Service Provision to Implement the World Health Organization HEARTS-D Guidelines in Bangladesh for Improving Diabetes Control and Prevention (HEARTS-D for Bangladesh)
Brief Title: Implementing WHO HEARTS-D Guidelines in Bangladesh for Diabetes Control and Prevention
Acronym: T2D IR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Projahnmo Research Foundation (Other); Johns Hopkins Bloomberg School of Public Health (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 115232; 1R01HL175636-01 (NIH)
Record Dates: First submitted 2025-07-10; First posted 2025-09-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes (T2DM)
Keywords: T2D IR; HEARTS-D; Type 2 Diabetes; Implementation Research; Non-communicable disease (NCD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, type-2 hybrid effectiveness-implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The community-to-facility integrated strategy (Experimental): The community-to-facility integrated strategy arm will focus on a joined-up T2D care delivery across the primary, secondary, and healthcare facilities, and urban communities. The intervention arm includes community-based care where Community Health Workers (CHWs) visit households to identify eligible individuals and refer them to relevant facilities. This arm will involve (i) 10 randomly chosen ward clusters, and (ii) primary health care centers and Community Health Workers (CHWs) serving these wards.
  Interventions: Other: The community-to-facility integrated strategy
- Existing services with no additional involvement of the PHCC-based CHWs (No Intervention): The remaining 10 ward clusters not included in the intervention arm will be considered as the comparison arm. The participants in this arm will receive the existing conventional services for diabetes in the PHCC and other clinical facilities. However, unlike the experimental arm, there will be no additional involvement of the PHCC-based CHWs in community-based screening and referral.

INTERVENTIONS:
Other: The community-to-facility integrated strategy — The community-to-facility integrated strategy will focus on a joined-up T2D care delivery across the primary, secondary, and healthcare facilities, and urban communities.
  Arms: The community-to-facility integrated strategy

SUMMARY:
Type-2 diabetes (T2D) is rising at an alarming rate in the low- and middle-income countries (LMIC). This rapid increase in the T2D burden has a particular impact on cities, where more than half the LMIC populations currently live and where 3 out of 4 people with T2D reside. In response to this growing global challenge, the World Health Organization (WHO) has emphasized (a) the need for an equitable and sustained improvement in the detection, treatment, and control of T2D, and (b) a rapid implementation of the WHO's evidence-based HEARTS-D module. However, currently, in most LMICs (such as Bangladesh), effective adoption of the WHO HEARTS-D module into routine urban primary care has been limited. These include suboptimal delivery mechanisms, poor uptake, weak monitoring system, and inadequate capacities. To address this, the investigators will evaluate a community-to-facility integrated strategy to implement WHO HEARTS-D module in the existing urban service delivery system in Bangladesh. First, the investigators will develop and optimize a community-to-facility integrated strategy for adopting the WHO HEARTS-D module using Implementation Mapping. Guided by this approach, the investigators will conduct mixed methods assessments to: (a) identify contextual factors, and (b) assess the implementation behavior of providers that may influence T2D care in cities. The investigators will then develop and optimize a suitable implementation strategy that can achieve high coverage, access and utilization of T2D care, specifically for urban poor populations, through iterative cycles of mixed methods qualitative assessments, implementation, and outcome measurements. For this aim, study staff will select the key stakeholders, primary care providers and CHWs as participants, based in 3 wards in Sylhet city of Bangladesh. Second, the investigators will evaluate the impacts of the optimized community-to-facility integrated strategy on implementation outcomes. The investigators will conduct a 2-arm, type 2, hybrid implementation-effectiveness randomized trial. The study will involve 20 municipal wards as clusters from Sylhet city (10 in each arm). This study compare the following strategies: (a) a community-to-facility integrated strategy for implementing the WHO HEARTS-D module and (b) a facility-only usual service delivery. The investigators will evaluate the implementation process by relevant outcomes based on the RE-AIM framework components: reach, effectiveness, implementation, and maintenance. Third, the investigators will compare the effectiveness of this strategy on T2D status. In a study sample of 10,000 randomly selected participants, the investigators will compare improvements in the prevalence of controlled T2D, treatment uptake and adherence to glucose-lowering therapy, T2D complications and awareness among participants in both study arms from baseline to end-line. Our study should guide the policymakers into effective implementation and sustainment of WHO HEARTS-D module that can be: (a) embedded within local organizational structures, and (b) adapted to similar contexts globally.

DETAILED DESCRIPTION:
Background Type-2 diabetes (T2D) is rising at an alarming rate in all low- and middle-income countries (LMIC). This rapid acceleration of the T2D burden has a particular impact on cities, where more than half the LMIC populations currently live and where 3 out of 4 people with T2D reside. In response to this growing global challenge, the World Health Organization (WHO) has emphasized the rapid implementation of the WHO's evidence-based HEARTS-Diabetes (HEARTS-D) module in all member states, which aims to improve service delivery for T2D in primary care facilities using highly effective, scalable, and proven strategies.

Currently, in most LMICs, effective adoption of the WHO HEARTS-D module into routine urban primary care has been limited owing to substantial implementation barriers. This also underscores a global unmet need for implementation research, which could help develop strategies to integrate and sustain this evidence-based module into practice. The Government of Bangladesh committed to rolling out the WHO HEARTS-D module as well. However, like the majority of LMICs, it faces implementation challenges regarding an effective strategy to adopt this module - owing to a lack of relevant implementation research data.

Aims and objectives This implementation research study aims to develop an optimized community-to-facility implementation model to strengthen urban healthcare for T2D management in Bangladesh using the WHO HEARTS-D module. The study will also evaluate the optimized implementation model to investigate its impact and effectiveness on T2D care in an urban setting in Bangladesh.

Study design This is an implementation research study, which will use a mixed-methods design, including both qualitative and quantitative research methodologies.

First, a formative research method will be used to identify barriers and facilitators for community-to-facility WHO HEARTS-D module implementation to design and optimize the initial implementation model. Concurrent program learning using qualitative research and outcome measurement while implementing the initial model in routine care settings will be used to improve the model iteratively until a high coverage of T2D care using the WHO HEARTS-D module is achieved. This process will produce the final, optimized WHO HEARTS-D implementation model, developed from the perspective of sustainable scale-up.

Second, the optimized implementation model will be evaluated by a type-2, hybrid implementation/effectiveness cluster-randomized trial. This trial will evaluate the program implementation and effectiveness of the final optimized model. For evaluating the implementation outcomes, the program elements for sustainable adoption and implementation of the integrated strategy will be assessed using the RE-AIM framework. For evaluation of effectiveness outcomes, data will be collected from a randomly selected study sample of 5000 individuals (i.e., samples included in the baseline and end-line survey).

Study setting The study will be conducted in the Sylhet City Corporation, Sylhet. During the development of the optimized model, three wards of the Sylhet City Corporation will be utilized. During the cluster randomized trial, 20 randomly selected wards will be utilized excluding the three wards which will be used for model development.

Study population For the implementation model optimization and evaluation, the community study population will include any individuals, who are ≥35 years of age and at risk of developing T2D, living in the study area. Additionally, the study will also include participants from the healthcare facilities including healthcare providers and community stakeholders relevant to local T2D care (e.g., local physicians, non-physician health workers, community health workers, and local community leaders) to conduct the qualitative research components of the study.

Study outputs and outcomes The main output of the first phase of this research project is to iteratively develop an optimized implementation model that achieves high coverage of T2D care in Sylhet City using the WHO HEARTS-D module. The performance of this optimized implementation model will then be evaluated through the implementation and effectiveness measures. The investigators will evaluate the implementation process by defining relevant outcomes based on the RE-AIM framework components: reach, effectiveness, implementation, and maintenance (e.g., intervention costs). The effectiveness outcomes will include the prevalence of controlled T2D status, treatment uptake and adherence to glucose-lowering therapy, T2D complications, and awareness among participants in both study arms, from baseline to end-line.

ELIGIBILITY:
Inclusion Criteria:

1. Adult individuals, ≥35 years of age,
2. Of either sex,
3. Long-term residents in the study area (defined by being a homeowner or a resident for at least the past three years), and
4. Willing to provide informed consent for study procedures and follow-up.

Exclusion Criteria:

1. Individuals planning to migrate from the study area before completing the first 12-month follow-up period, and
2. Individuals explicitly requesting exclusion from the study or unable to provide consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Implementation of the Community-to-Facility Integrated Care Intervention | Baseline; and through study completion, an average of 1 year.
  This outcome will measure the extent to which the integrated community-to-facility care intervention has been successfully implemented, based on the RE-AIM framework.
Effectiveness of the Community-to-Facility Integrated Care Intervention on Health Outcome | Baseline; and through study completion, an average of 1 year
  This outcome will evaluate the effectiveness of the intervention by measuring the percentage of study participants with uncontrolled T2D

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah H Baqui, DrPH, Study Chair — Johns Hopkins Bloomberg School of Public Health

IPD SHARING:
Plan to Share IPD: Yes